CLINICAL TRIAL: NCT06315309
Title: Phase II Clinical Trial of 2 Step ATG Combined With Tacrolimus and Mini Methotrexate for Prevention of Acute GVHD Post Myeloablative Allogeneic Stem Cell Transplant
Brief Title: Trial of 2 Step ATG for Acute GVHD Prevention Post Myeloablative Allogeneic Stem Cell Transplant
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Zaid Al-Kadhimi, Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300012281 (UAB 23146); Robert Award (Other: University of Alabama at Birmingham)
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: GVHD,Acute; Acute Leukemia; Myelodysplastic Syndromes; Myeloproliferative Disorders
Keywords: Leukemia; Myelodysplastic Syndrome; Myeloproliferative Disorders
MeSH Terms: conditions — Myelodysplastic Syndromes; Myeloproliferative Disorders; Leukemia | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- phase II single arm study of 2 step ATG dosing in prevention of aGVHD. (Experimental): The primary outcome for the study is rate of GRFS at one-year post transplant. When accounting for competing risks, any death, relapse, Grade III-IV acute GVHD and cGVHD requiring systemic therapy are competing risks. The reported one year GRFS with the use of standard of care GVHD prevention regimen in MA HSCT (Tac/MTX) was 35%. (El-Jurdi 2023) We hypothesize that with 2 step ATG/Tac/Mini MTX regimen, we can achieve a one year GRFS of 60%.
  Interventions: Drug: ATG Combined with Tacrolimus and Mini Methotrexate

INTERVENTIONS:
Drug: ATG Combined with Tacrolimus and Mini Methotrexate — On Day -7, subjects will be admitted to the hospital and receive a dose of prednisone at 1 mg/kg (ATG premedication). Subjects will receive a steroid injection 3 hours before every ATG infusion. On day -6, subjects will receive a small dose of ATG as an IV infusion. ATG will be repeated on days -5,-4 and -1. Routine transplant chemotherapy agent fludarabine will be given on days -6 to -2 as daily IV infusions. Busulfan, a routine transplant chemotherapy will be given on days -5 to -2 as IV infusion. Subjects with lymphoblastic leukemia will receive an alternative regimen of cyclophosphamide, a routine chemotherapy on days -6 and -5, followed by total body radiation on days -3 to -1. Tacrolimus (standard immune suppression agent) starts on day -3 as continuous IV infusion and switched to oral after engraftment. Methotrexate a standard immune suppression medication which is given IV on day +1,+3,+6, and +11 post-transplant. Blood draws on days -4,-1,+3,+7,+14 to measure ATG levels.

SUMMARY:
The purpose of this study is to test whether the combination of the drugs called tacrolimus (Tac), methotrexate (MTX) and new dosing strategy of another drug called (rabbit Anti-thymocyte Globulin [ATG]) will help prevent the development and/or improve severity of acute and/or chronic GVHD.

DETAILED DESCRIPTION:
The goal is to study the effectiveness and drug levels of new dosing strategy of ATG (GVHD preventing medicine) in preventing graft versus host disease post allogeneic stem cell transplantation.

In an effort to reduce graft versus host disease (GVHD) and enhance graft versus leukemia (GVL) effect post allogenic hematopoietic stem cell transplantation (AHSCT), recent research has focused on host immune cell depletion. Frame shifting anti-thymocyte globulin (ATG) backwards to earlier days before days 0 can result in deeper host and less graft T-cell depletion, leading to better immune reconstitution. Preliminary data where 80% of the ATG dose is given on days -6,-5,-4 and 20% given on day -1, showed effective prevention of severe acute GVHD, chronic GVHD and favorable early immune reconstitution. We hypothesize that our 2 step ATG dosing platform when combined with standard tacrolimus and mini methotrexate in a myeloablative setting can prevent grade III-IV acute GVHD and chronic GVHD, resulting in improvement of GVHD/relapse free survival at one year post transplant.

This study aims to:

1. Confirm the effectiveness of ATG based GVHD prevention regimen based on the encouraging clinical outcomes observed above.
2. Examine ATG blood levels pre and post-transplant to evaluate any possible correlation between ATG levels and its ability to protect from GVHD.
3. Examine post-transplant immune cell recovery as part of routine post-transplant immune monitoring at UABMC.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female, age 18-60 years
2. Patients must have a related or unrelated peripheral blood stem cell donor. Sibling donor must be a 6/6 match for HLA-A and -B at intermediate (or higher) resolution, and -DRB1 at high resolution using DNA-based typing, and must be willing to donate peripheral blood stem cells and meet institutional criteria for donation. Unrelated donor must be 8/8 match at HLA-A, -B, -C and -DRB1 at high resolution using DNA-based typing. Unrelated donor must be willing to donate peripheral blood stem cells and be medically eligible to donate stem cells according to NMDP criteria.
3. A candidate for Myeloablative preparative regimen, based on age ≤ 60, or HCT-CI of ≤ 4, and considered by the treating physician to be a candidate for such regimen.
4. Cardiac function: Ejection fraction ≥ 45%
5. Calculated creatinine clearance greater than 50 mL/minute (using the Cockcroft-Gault formula and actual body weight).
6. Pulmonary function: DLCO ≥50% (adjusted for hemoglobin) and FEV1≥50%
7. Liver function: total bilirubin < 1.5x the upper limit of normal and ALT/AST < 2.5x the upper normal limit. Patients who have been diagnosed with Gilbert's Disease are allowed to exceed the defined bilirubin value up to <3mg/dl.
8. Female subjects (unless postmenopausal for at least 1 year before the screening visit, or surgically sterilized), agree to practice two effective methods of contraception (hormonal contraception and male partner to use condom) or agree to complete abstain from heterosexual intercourse from the time of signing the informed consent through 12 months post-transplant.
9. Male subjects (even if surgically sterilized), of partners of women of childbearing potential must agree to practice effective barrier contraception or abstain from heterosexual intercourse from the time of signing the informed consent through 12 months post-transplant.
10. Karnofsky performance status KPS ≥ 80 (Appendix B)
11. Patients must have a diagnosis of one of the following:

    A-Acute myeloid leukemia (AML) in complete remission CR 1 with intermediate or high risk for relapse as defined by ELN 2022 criteria(Dohner et al., 2022) (appendix C), or deemed to be at high risk for relapse by treating physician, based on, therapy related, or extra medullary presentation.

    B-AML in >CR1. C-Myelodysplastic syndrome (MDS) with IPSS-M ≥ intermediate-low.(Bernard et al., 2022; Mohty et al., 2022) D- Chronic myeloproliferative disorder (ET, PV, myelofibrosis) with bone marrow blasts > 5% and/or other evidence of progression to acute leukemia or Int or high-risk disease by MIPPS v2 score.(Ali et al., 2019; Guglielmelli et al., 2018) E- CMML especially those with high-risk features based in: The CMML-specific prognostic scoring system with molecular features (CPSS-Mol) - high risk and intermediate-2 risk, Mayo molecular model - high risk and Intermediate-2 risk, Groupe Francophone des Myélodysplasies (GFM) - high risk and selected patients with intermediate risk.(Elena et al., 2016; Itzykson et al., 2013; Patnaik et al., 2014). F- Acute lymphoblastic leukemia (ALL) in CR1 with high risk for relapse
    * B-cell ALL: High white blood cell count at diagnosis (ie, >30,000/µl), Clonalcytogenetic abnormalities - t(4;11), t(1;19), t(9;22), or BCR-ABL gene positivity, BCR-ABL1-like (Ph-like) gene signature, progenitor-B cell immunophenotype (eg, blasts expressing membrane CD19, CD79a, and cytoplasmic CD22, but not CD10), Length of time from start of induction therapy to attainment of CR greater than four weeks, and minimal residual disease (MRD) post-remission bone marrow MRD+.(Akabane & Logan, 2020; Lafage-Pochitaloff et al., 2017)
    * T-cell ALL: Failure to achieve CR after one induction, MRD> 1X 10-4 after 2 courses of induction, Presenting WBC > 100 X 109/L, complex cytogenetics ≥5,early T-cell Precursor ALL, poor risk genetics including lack of NOTCH1 ith/FBXW7 or presence of N-RAS & K-RAS, EZH2 and age>40 years.(Marks & Rowntree, 2017) G- ALL in >CR1
12. The subject is willing and able to sign informed consent and abide by the protocol requirements.

Exclusion Criteria:

1. Autologous hematopoietic stem cell transplant < 3 months prior to enrollment.
2. Patients with florid residual AML with > 5% blast in the marrow or circulating blast in the peripheral blood are not eligible for this study.
3. Previous allogeneic stem cell transplant.
4. Uncontrolled angina, severe uncontrolled ventricular arrhythmias, or EKG suggestive of acute ischemia or active conduction system abnormalities.
5. Known hypersensitivity to the study agent (ATG)
6. Received any investigational drugs within the 14 days prior to the first day of transplant conditioning
7. Pregnant and/or breastfeeding
8. Evidence of HIV infection or known HIV positive serology.
9. Current uncontrolled bacterial, viral or fungal infection (currently taking medication with evidence of progression of clinical symptoms or radiologic findings).
10. Non-hematologic malignancy within prior three (3) years, with the exception of squamous cell or basal cell skin carcinoma.
11. Participation in another clinical study with an investigational product during the last 28 days.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
To estimate the therapeutic success of 2-step ATG dosing platform in patients undergoing reduced intensity allogeneic transplantation for treatment of hematologic malignances | 1 year post transplant
  Rate of GRFS (graft versus host disease GVHD, relapse free survival) at one year post transplant. To meet that end point the patient needs to be alive without relapse, or grade III-IV acute GVHD, or chronic GVHD requiring systemic immune suppression.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States